CLINICAL TRIAL: NCT03108755
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP7713 in Healthy Non-Japanese Adult and Elderly Subjects and Healthy Japanese Adult Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP7713 in Healthy Non-Japanese Adult and Elderly Subjects and Healthy Japanese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 7713-CL-0001; 2016-004845-10 (EudraCT Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: ASP7713

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ASP7713 Single Ascending Dose (Experimental): Successive cohorts of 8 non-Japanese participants (6 ASP7713/ 2 Placebo / 1-7 cohorts) will be started on a fixed single dose of ASP7713 or matching Placebo. The first two participants will receive either ASP7713 or matching placebo. If no safety issues are observed in the first 24 hours in the first two participants, then the remaining six participants will be dosed. Safety, tolerability and available Pharmacokinetic data from proceeding cohorts will be assessed for dose escalation.
  Interventions: Drug: ASP7713
- Placebo Single Ascending Dose (Placebo Comparator): Successive cohorts of 8 non-Japanese participants (6 ASP7713/ 2 Placebo / 1-7 cohorts) will each be started on a single fixed dose of ASP7713 or matching Placebo. The first two participants will receive either ASP7713 or matching placebo. If no safety issues are observed in the first 24 hours in the first two participants, then the remaining six participants will be dosed. Safety, tolerability and available Pharmacokinetic data from proceeding cohorts will be assessed for dose escalation.
  Interventions: Drug: Placebo
- ASP7713 Multiple Ascending Dose (Adults: 18-55 years) (Experimental): Successive cohorts of 16 participants consisting of 8 non-Japanese and 8 Japanese (12 ASP7713/ 4 Placebo /1-3 cohorts) will each be started on a fixed multiple dose of ASP7713 or matching Placebo twice or three times daily for 14 days. Safety, tolerability and available Pharmacokinetic data from proceeding cohorts will be assessed for dose escalation.
  Interventions: Drug: ASP7713
- Placebo Multiple Ascending Dose (Adults: 18-55 years) (Placebo Comparator): Successive cohorts of 16 participants consisting of 8 non-Japanese and 8 Japanese (12 ASP7713/ 4 Placebo /1-3 cohorts) will each be started on a fixed multiple dose of ASP7713 or matching Placebo twice or three times daily for 14 days. Safety, tolerability and available Pharmacokinetic data from proceeding cohorts will be assessed for dose escalation.
  Interventions: Drug: Placebo
- ASP7713 Multiple Ascending Dose (Elderly: 65 years or older) (Experimental): Dosing of the non-Japanese elderly cohort will commence after having established the safety and tolerability of corresponding dose in adults male and female participants.
  Interventions: Drug: ASP7713
- Placebo Multiple Ascending Dose (Elderly: 65 years or older) (Placebo Comparator): Dosing of the non-Japanese elderly cohort will commence after having established the safety and tolerability of corresponding dose in adults male and female participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7713 — oral
  Arms: ASP7713 Multiple Ascending Dose (Adults: 18-55 years); ASP7713 Multiple Ascending Dose (Elderly: 65 years or older); ASP7713 Single Ascending Dose
Drug: Placebo — oral
  Arms: Placebo Multiple Ascending Dose (Adults: 18-55 years); Placebo Multiple Ascending Dose (Elderly: 65 years or older); Placebo Single Ascending Dose

SUMMARY:
This is a combined Single and Multiple Ascending Oral Dose Study. Part 1 is a Single Ascending Dose (SAD) and Part 2 is Multiple Ascending Dose (MAD).

The purpose of the study is to evaluate the safety and tolerability of single and multiple ascending oral doses of ASP7713 in healthy non-Japanese (Part 1) and Japanese (Part 2) adult participants and non-Japanese elderly participants (Part 2).

This study will also evaluate the pharmacokinetics of single and multiple ascending oral doses of ASP7713 in non-Japanese (Part1) and Japanese (Part 2) adult participants and non-Japanese elderly participants (Part 2) as well as the effect of a single and multiple oral dose of ASP7713 on the QT interval using Fridericia's Correction (QTcF).

In addition, this study will evaluate a potential racial difference in safety, tolerability and pharmacokinetics of multiple oral doses of ASP7713 in healthy non-Japanese and Japanese adult participants (Part 2).

DETAILED DESCRIPTION:
There will be a residential period for Parts 1 and 2. Part 1: Eligible participants will be residential for a single period of 5 days and 4 nights. Participants will be discharged on day 4 on the condition that all required assessments have been performed and that there are no medical reason for a longer stay in the clinical unit.

Part 2: Eligible participants will be residential for a single period of 18 days and 17 nights. Participants will be discharged on day 17 on the condition that there are no medical reason for a longer stay in the clinical unit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy non-Japanese adult male or female subject between 18 to 55 years of age, inclusive, at screening or subject is a healthy non-Japanese elderly male or female subject, ≥ 65 years of age and has a body mass index (BMI) range of 18.5 to 30.0 kg/m2, inclusive and weighs at least 50 kg at screening and day -1 OR Subject is a healthy Japanese adult male or female subject between 20 to 55 years of age, inclusive, at screening and has a BMI range of 18.0 to 28.0 kg/m2, inclusive and weighs at least 45 kg at screening and day -1.
* In case of Japanese subject: subject is from Japanese origin. Both parents and all 4 grandparents should be Japanese. The subject should have been born in Japan and should not have lived outside of Japan for more than 10 years.
* Female subject must either:

  * Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses) prior to screening, or Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) Or, if of childbearing potential, Agree not to try to become pregnant during the study and for 28 days after the final study drug administration, And have a negative pregnancy test at day -1, And if heterosexually active, agree to consistently use 2 forms of birth control (1 of which is a highly effective method and 1 must be a barrier method) starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * Male subject agrees to use a male condom starting at screening and continue throughout study treatment and for 28 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a male condom for the duration of the pregnancy or for the time the partner is breastfeeding throughout the study period and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received investigational therapy within 28 days (or 5 half-lives, whichever is longer) prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP7713, or any components of the formulation used.
* Subject has had previous exposure with ASP7713.
* Subject has any of the liver function tests (LFTs) (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma-glutamyl transferase and total bilirubin [TBL]) above the upper limit of normal (ULN) at day -1. In such a case, the assessment may be repeated once.
* Subject has any of the cardiac troponins (cardiac troponin T [cTnT] and cardiac troponin I [cTnI]) above the ULN at day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG) and protocol-defined safety laboratory tests at screening or day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure < 90 or > 140 mmHg; mean diastolic blood pressure < 50 or > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) at screening or day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean QTcF interval of > 430 msec (for males) and > 450 msec (for females) at screening or day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of long QT syndrome.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day) and except for use of hormonal contraceptives and hormone replacement therapy.
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past 6 months prior to screening.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14 units of alcohol for female subjects) within 3 months prior to day -1 or the subject tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 3 months prior to day -1.
* Subject has consumed grapefruit/Seville oranges, grapefruit-containing products or Seville orange-containing products within 72 hours prior to admission to the clinical unit.
* Subject has used any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibody, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of the Astellas Group or contract research organization.
* Subject has a history of orthostatic hypotension or a positive orthostatic challenge test which is based on the measurements 3 minutes after standing:

  * Systolic blood pressure (SBP) ≥ 20 mmHg decrease from supine and/or
  * Diastolic blood pressure (DBP) ≥ 10 mmHg decrease from supine at screening or day -1.
* Subject has any clinically significant abnormalities on cardiac imaging at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by nature, frequency and severity of Adverse Events (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Treatment Emergent Adverse Event (TEAE) is defined as any AE starting or worsening at any time from first dosing until last scheduled procedure.
Number of Participants with Vital Sign Abnormalities and/or Adverse Events (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with Laboratory Value Abnormalities and/or Adverse Events (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Number of participants with potentially clinically significant laboratory values.
Safety assessed by routine 12-Lead Electrocardiogram (ECG) (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Any clinically significant adverse changes on the ECG will be reported as an AE.
Safety assessed by continuous 12-Lead Electrocardiogram (ECG) (Part 1 and Part 2) | Part 1: Up to Day 2 / Part 2: Up to Day 17
  Any clinically significant adverse changes on the ECG will be reported as an AE.
Safety assessed by Real-time cardiac monitoring (telemetry) (Part 1) | Part 1: Up to Day 1
  Number of participants with potentially clinically significant telemetry abnormalities.
Safety assessed by Cardiac troponin T (cTnT) (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Number of participants with potentially clinically significant cTnT abnormalities. Cardiac troponin T is a component of the contractile apparatus of myocardial cells and is expressed almost exclusively in the heart.
Safety assessed by Cardiac troponin I (cTnI) (Part 1 and Part 2) | Part 1: Up to Day 16 / Part 2: Up to Day 29
  Number of participants with potentially clinically significant cTnI abnormalities. Cardiac troponin I is a component of the contractile apparatus of myocardial cells and is expressed almost exclusively in the heart.
Safety assessed by Orthostatic challenge test (OCT) (Part 1 and Part 2) | Part 1: Up to Day 1 / Part 2: Up to Day 14
  Number of participants with potentially clinically significant OCT changes will be reported as an AE.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) of ASP7713 in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 7
  AUCinf will be derived from the pharmacokinetic (PK) plasma samples collected.
Part 1: PK of ASP7713 in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to Day 7
  AUClast will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: percentage of AUCinf due to extrapolation from time of the last measurable concentration to time infinity (AUCinf(%extrap)) | Up to Day 7
  AUCinf(%extrap) will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: maximum concentration (Cmax) | Up to Day 7
  Cmax will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: apparent total systemic clearance after extravascular dosing (CL/F) | Up to Day 7
  CL/F will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: time prior to the time corresponding to the first measurable (nonzero) concentration (tlag) | Up to Day 7
  tlag will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: time of maximum concentration (tmax) | Up to Day 7
  tmax will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: terminal elimination half-life (t ½) | Up to Day 7
  t ½ will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in plasma: apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F) | Up to Day 7
  Vz/F will be derived from the PK plasma samples collected.
Part 1: PK of ASP7713 in urine: cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast) | Up to Day 4
  Aelast will be derived from the PK urine samples collected.
Part 1: PK of ASP7713 in urine: percentage of study drug dose excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast%) | Up to Day 4
  Aelast% will be derived from the PK urine samples collected.
Part 1: PK of ASP7713 in urine: cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf) | Up to Day 4
  Aeinf will be derived from the PK urine samples collected.
Part 1: PK of ASP7713 in urine: percentage of study drug dose excreted into urine from time of dosing extrapolated to time infinity (Aeinf%) | Up to Day 4
  Aeinf% will be derived from the PK urine samples collected.
Part 1: PK of ASP7713 in urine: renal clearance (CLR) | Up to Day 4
  CLR will be derived from the PK urine samples collected.
Part 2: PK of ASP7713 in plasma: area under the concentration-time curve from the time of dosing to 24 hours postdose (AUC24) | Day 1
  AUC24 will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: area under the concentration-time curve from the time of dosing to 12 hours postdose (AUC12) | Days 1 and 14
  AUC12 will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: area under the concentration-time curve from the time of dosing to 8 hours postdose (AUC8) | Days 1 and 14
  AUC8 will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: Cmax | Day 1, Day 12 (for twice daily dosing) and Day 14
  Cmax will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: tlag | Day 1
  tlag will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: tmax | Day 1, Day 12 (for twice daily dosing) and Day 14
  tmax will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau) | Day 12 (for twice daily dosing) and Day 14
  AUCtau will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: apparent total systemic clearance after extravascular dosing (CL/F) | Day 12 (for twice daily dosing) and Day 14
  CL/F will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: peak trough ratio (PTR) | Day 12 (for twice daily dosing) and Day 14
  PTR will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: accumulation ratio calculated using the area under the concentration time (Rac(AUC)) | Day 12 (for twice daily dosing) and Day 14
  Rac(AUC) will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: t ½ | Day 12 (for twice daily dosing)
  t ½ will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in plasma: Vz/F | Day 12 (for twice daily dosing)
  Vz/F will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in urine: cumulative amount of study drug excreted into urine from the time of dosing to the start of the next dosing interval (Aetau) | Day 14
  Aetau will be derived from the PK urine samples collected.
Part 2: PK of ASP7713 in urine: percentage of study drug dose excreted into urine from the time of dosing to the start of the next dosing interval (Aetau%) | Day 14
  Aetau% will be derived from the PK urine samples collected.
Part 2: PK of ASP7713 in urine: CLR | Day 14
  CLR will be derived from the PK urine samples collected.
Part 2: PK of ASP7713 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Days 2, 4, 6, 8, 10, 12 (for twice or 3 times daily dosing) , 14 and 15
  Ctrough will be derived from the PK plasma samples collected.
Part 2: PK of ASP7713 in urine: concentration immediately prior to dosing at multiple dosing (Ctrough) | Days 2, 4, 6, 8, 10, 12 (for twice or 3 times daily dosing), 14 and 15
  Ctrough will be derived from the PK urine samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site GB44001, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided